CLINICAL TRIAL: NCT01339143
Title: An Open-label, Randomized, Active-controlled Study to Compare the Effect of DPP-IV Inhibitor and TZD as add-on Therapy to Metformin on Glycemic Variability and Oxidative Stress in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy
Brief Title: Compare the Effect of DPP-IV Inhibitor or TZD on Glycemic Variability and Oxidative Stress in Patient With 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Sin-Gon Kim, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN10016-002
Record Dates: First submitted 2011-04-15; First posted 2011-04-20 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2010-04

CONDITIONS: Diabetes Mellitus; Oxidative Stress
Keywords: Vildagliptin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vildagliptin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Active Comparator): pioglitazone: 15mg, QD, PO, 16 weeks
  Interventions: Drug: pioglitazone
- vildagliptin (Experimental): vildagliptin 50mg,BID,PO,16 weeks
  Interventions: Drug: Galvus (vildagliptin)

INTERVENTIONS:
Drug: Galvus (vildagliptin) — 50mg BID, PO, for 16 weeks
  Arms: vildagliptin
Drug: pioglitazone — 15mg, QD, PO, 16 weeks
  Arms: Pioglitazone

SUMMARY:
The purpose of this study is to compare the effect of vildagliptin vs. pioglitazone to oxidative stress on daily blood glucose fluctuations, in patients with type 2 diabetes that was inadequately controlled by metformin.

DETAILED DESCRIPTION:
Activation of oxidative stress by glucose fluctuations plays a major role in the pathogenesis of diabetic complication. Dipeptidyl peptidase IV (DPP-IV), such as vildagliptin, enhances glucose-induced insulin secretion, decreases glucagon secretion, and reduces postprandial hyperglycemia and may also improve acute fluctuations of glucose. We believe that vildagliptin may exert an effect of decreasing oxidative stress by reducing glucose excursion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with age 18-80 years
* Type 2 diabetes mellitus
* On stable dose of metformin (more than 1000mg) for at least 1 month
* HbA1c 7~10%
* Subjects on statins, ACE inhibitors, ARBs and antioxidants will be allowed as long as they are on stable doses of these compounds and the dosage is not changed during the course of study
* BP under control - no change required to BP medications
* Agreement to maintain prior diet & exercise

Exclusion Criteria:

* Type 1 DM or Any kind of secondary DM
* Pregnant or lactating women.
* Treatment with sulfonylurea, α-glucosidase inhibitor, glinide, GLP-1 analogues, DPP-IV inhibitors or insulin therapy within 1 month prior to informed consent.
* Treatment with rosiglitazone or pioglitazone within 3 months prior to informed consent.
* HbA1c <7% or >10%
* Uncontrolled hypertension ( BP > 160/100 mmHg)
* Congestive heart failure (NYHA class I to IV).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Glycemic Variability | 16 weeks

SECONDARY OUTCOMES:
Oxidative stress | 16 weeks
HbA1C | 16 weeks
hypoglycemia | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea